CLINICAL TRIAL: NCT06673979
Title: Risk Factors Affecting Chronic Postoperative Pain After Elective Nephrectomy
Brief Title: Risk Factors for Chronic Postoperative Pain After Elective Nephrectomy
Status: Recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, İlayda Bilgili Altuntaş, Principal investigator, Anesthesiology and Reanimation, Physician, Istanbul University - Cerrahpasa
Other Study IDs: E-83045809-604.01-1084787
Record Dates: First submitted 2024-09-25; First posted 2024-11-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: General Anesthesia; Chronic Pain, Postoperative; Acute Pain, Postoperative; Surgery; Anesthesia; Chronic Pain; Analgesic Drugs; Epidural Analgesia; Nephrectomy
Keywords: chronic pain; nephrectomy; surgery; pain risk factors; acute pain; postoperative pain
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain; Acute Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Painfull: patients with Numeric Rating Score equal or higher than 4: The patients are asked to rate their pain according to the Numeric Rating Scale (0=no pain; 10=worse possible pain), and patients with NRS equal or higher than 4 are defined as "painfull".
  Interventions: Diagnostic Test: Numeric Rating Scale
- Pain-free: patients with Numeric Rating Score lower than 4: The patients are asked to rate their pain according to the Numeric Rating Scale (0=no pain; 10=worse possible pain), and patients with NRS lower than 4 are defined as "pain-free".
  Interventions: Diagnostic Test: Numeric Rating Scale

INTERVENTIONS:
Diagnostic Test: Numeric Rating Scale — The patients are asked to rate their pain according to the Numeric Rating Scale (0=no pain; 10=worse possible pain).

SUMMARY:
Chronic postoperative pain (CPP) is typically defined as pain persisting for 3 months or more after surgery[1]. CPP is a common and increasingly prevalent morbidity, leading to long-term psychological issues, reduced quality of life, and impaired functionality[2]. To reduce the incidence of CPP, high-risk patients are identified, and various surgical techniques, pharmacological agents, and regional anesthesia techniques are employed[3].

The primary aim of our study is to scale chronic pain at 1 hour, 3 months, and 1 year post-nephrectomy using the Numeric Rating Scale (NRS), ranging from 0 to 10. The secondary aim is to evaluate the effects of factors influencing chronic postoperative pain on the NRS scores.

DETAILED DESCRIPTION:
Patients gender, age, height(m), weight(kg), body mass index(kg/m2), diagnosis, smoking and alcohol history, comorbidities, surgical technique and duration, complications, lymph node dissection, thrombectomy, adrenalectomy, amount of bleeding(cc), need for blood transfusion, need for intensive care, analgesia technique used, amount of opioids and non-opioid analgesics used perioperatively, amount of vasopressors used, heart rate(bpm) and mean arterial pressure(mmHg) at induction, post-intubation, post-extubation, and 1 hour postoperatively, presence of postoperative pain, chronic analgesic use history(more than 3 uses per week), presence of fibromyalgia, frequent urinary tract infections, diagnosed with central sensitization disorders, bruxism, depression-panic attacks, allergic asthma, irritable bowel syndrome, and migraines will be recorded. The effects of these factors on NRS scores at 1 hour, 3 months, and 1 year postoperatively will be examined.

ELIGIBILITY:
Inclusion Criteria: -Patients aged 18-90 years,

* ASA I-IV,
* undergoing elective nephrectomy under general anesthesia will be included in the study.

Exclusion Criteria:

* Patients who cannot be reached by phone and hose who die within the 1-year postoperative period will be excluded from the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-90 years, ASA I-IV, undergoing elective nephrectomy under general anesthesia will be included in the study.
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
NRS 1 hour | 1 hour after the end of the surgery
  The patients are asked to rate their pain according to the Numeric Rating Scale (0=no pain; 10=worse possible pain). Patients with NRS equal or higher than 4 are defined as painfull; and, patients with NRS lower than 4 are defined as pain-free
NRS 3 months | 3 months after the surgery
  The patients are asked to rate their pain according to the Numeric Rating Scale (0=no pain; 10=worse possible pain). Patients with NRS equal or higher than 4 are defined as painfull; and, patients with NRS lower than 4 are defined as pain-free
NRS 1 year | 1 year after the surgery
  The patients are asked to rate their pain according to the Numeric Rating Scale (0=no pain; 10=worse possible pain). Patients with NRS equal or higher than 4 are defined as painfull; and, patients with NRS lower than 4 are defined as pain-free

SECONDARY OUTCOMES:
age | At the time of preoperative assesment
  Age of the patiens as years
height | At the time of preoperative assesment
  Height of the patiens as meter
BMI | At the time of preoperative assesment
  body mass index of the patiens as kg/m2
smoking | At the time of preoperative assesment
  Data of the patient if they are smoking or not
Amount of opioid and non-opioid analgesics used perioperatively | At the time of perioperative assesment
  Amount of opioid and non-opioid analgesics used perioperatively
Gender | At the time of preoperative assesment
  Woman or man
Comorbidities | At the time of preoperative assesment
  hipertension, diabetus mellitus, asthma or cardiac disease etc.
surgical technique | At the time of perioperative assesment
  radical or partial nephrectomy and open or laparoscopic nephrectomy
surgical duration | The time recorded at the end of the surgery will be reported
  How long does the surgery take in minutes?
additional procedures next to the nephrectomy | At the time of perioperative assesment
  lymph node dissection, thrombectomy, adrenalectomy procedures used
need for blood transfusion | At the time of perioperative assesment
  How many blood product tranfusions were required?
need for intensive care units | At the time of postoperative assesment, the data evaluated at the end of the surgery will be reported
  Whether there is a need for intensive care after surgery
Analgesia technique | At the time of perioperative assesment
  Epidural analgesia or intravenous analgesia was used as analgesic technique
Amount of vasopressors used | At the time of perioperative assesment
  Amount of vasopressors used at the perioperative period
Value of postoperative acute pain score on NRS score | 1 hour postoperative period
  Value of postoperative acute pain score on NRS score(0:no pain, 10:the worst pain imaginable)
Chronic analgesic use history | 1 year before the operation
  More than 3 uses per a week
Clinical conditions that will be reported under the title of central sensitization disorder | At the time of preoperative assesment
  Presence of fibromyalgia, frequent urinary tract infection, bruxism, diagnosed with depression-panic attack, allergic asthma, irritable bowel syndrome and migraines will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Aylin Nizamoglu, Doctor, Study Director — Istanbul Univerisity-Cerrahpasa Cerrahpasa Faculty of Medicine; Safak E Erbabacan, associate professor, Study Chair — Istanbul Univerisity-Cerrahpasa Cerrahpasa Faculty of Medicine; Fatis Altindas, Professor, Study Chair — Istanbul Univerisity-Cerrahpasa Cerrahpasa Faculty of Medicine; Ilayda Bilgili Altuntas, Physician, Principal Investigator — Istanbul Univerisity-Cerrahpasa Cerrahpasa Faculty of Medicine
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma LR, Schaldemose EL, Alaverdyan H, Nikolajsen L, Chen D, Bhanvadia S, Komen H, Yaeger L, Haroutounian S. Perioperative factors associated with persistent postsurgical pain after hysterectomy, cesarean section, prostatectomy, and donor nephrectomy: a systematic review and meta-analysis. Pain. 2022 Mar 1;163(3):425-435. doi: 10.1097/j.pain.0000000000002361. PMID 34121077
- See also: Perioperative factors associated with persistent postsurgical pain after hysterectomy, cesarean section, prostatectomy, and donor nephrectomy: A systematic review and meta-analysis — https://profiles.wustl.edu/en/publications/perioperative-factors-associated-with-persistent-postsurgical-pai